CLINICAL TRIAL: NCT01048541
Title: A Non-Inferiority Bladder Scan Study to Investigate Residual Urine After Use of Intermittent Catheters in Male Subjects
Brief Title: Bladder Scan of Residual Urine With New Catheter
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CP061CC
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SpeediCath catheter (Active Comparator): Standard treatment
  Interventions: Device: SpeediCath
- Test product (Experimental)
  Interventions: Device: Test Catheter - SpeediCath Compact Male

INTERVENTIONS:
Device: Test Catheter - SpeediCath Compact Male — Compact catheter for intermittent catheterisation
  Other Names: SpeediCath; Test catheter
  Arms: Test product
Device: SpeediCath — Catheter for intermittent catheterisation
  Other Names: Test catheter
  Arms: SpeediCath catheter

SUMMARY:
Male intermittent catheters (ICs) range from 340-500 mm long, with the European standard minimum length being 360 mm for a catheter without a balloon and 275 mm for one with a balloon. This length is defined by hospital standards although it is known that the male urethra has an approximate maximum length of 29 cmA new intermittent catheter developed by Coloplast A/S is a 30-cm-long sterile, ready-to-use, hydrophilic-coated male catheter. There is a lack of clinical data documenting that male ICs that are shorter and more or less flexible than standard catheters can sufficiently empty the bladder of male subjects. This will be tested using ultrasound to measure residual urine in the bladder following catheterisation with new product and standard length catheter.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male IC user able to self-catheterise
2. Subject has used hydrophilic-coated ICs for at least 1 month
3. Subject is at least 18 years old.
4. Subject has provided informed consent.

Exclusion Criteria:

1. Subject has symptoms of UTI (ie, fever, autonomic dysreflexia, spasticity, discomfort or pain over the kidney or bladder, onset/increase in incontinence episodes, cloudy urine with increased odour, malaise, lethargy, or sense of unease).
2. Subject has known abnormalities in the lower urinary tract.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Domurath, Dr. med., Principal Investigator — Werner Wicker Klinik; Henrik S Knoth, M.Sc Pharm, Study Director — Coloplast A/S
Locations (1):
- Werner-Wicker-Klinik, Abteilung für Neuro-Urologie, Bad Wildungen, Hesse, Germany

REFERENCES:
- [Derived] Prieto JA, Murphy CL, Stewart F, Fader M. Intermittent catheter techniques, strategies and designs for managing long-term bladder conditions. Cochrane Database Syst Rev. 2021 Oct 26;10(10):CD006008. doi: 10.1002/14651858.CD006008.pub5. PMID 34699062
- [Derived] Domurath B, Kutzenberger J, Kurze I, Knoth HS. Clinical evaluation of a newly developed catheter (SpeediCath Compact Male) in men with spinal cord injury: residual urine and user evaluation. Spinal Cord. 2011 Jul;49(7):817-21. doi: 10.1038/sc.2011.14. Epub 2011 Mar 1. PMID 21358718

RESULTS

PARTICIPANT FLOW:
Groups:
- AB: First Test Catheter Then Standard Catheter: Test catheter (SpeediCath Compact Male)used in the first period and Standard catheter (SpediCath straight) used in the second period
- BA: First Standard Catheter Then Test Catheter: Standard catheter (SpediCath straight)used in the first period and test catheter (SpeediCath Compact Male) used in the second period
Period: Overall Study
Arm/Group | AB: First Test Catheter Then Standard Catheter | BA: First Standard Catheter Then Test Catheter
Started | 18 | 19
Completed | 17 | 19
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study: Includes groups randomized to standard catheter first and test catheter first
Arm/Group | Entire Study
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 37
Region of Enrollment [Number; unit: participants]
  Germany | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Residual Urine Volume
Description: Residual urine was mesured by ultrasound measurement of bladder content after intermittent catherisation
Time Frame: 3 catheterisations on 1 day
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Test Catheter: Test catheter (SpeediCath Compact Male)
- Standard Catheter: Standard catheter (SpediCath straight)
Arm/Group | Test Catheter | Standard Catheter
Number analyzed (Participants) | 36 | 36
mL | 12.4 (15.7) | 9.4 (11.4)

2. Secondary Outcome: The Difference in Incidence of Adverse Events (AEs) and Adverse Device Events (ADEs)
Time Frame: Study period
Reporting Status: Not Posted

3. Secondary Outcome: Median Absolute RU Volume
Time Frame: 3 catheterisations on 1 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Test Catheter | Standard Catheter
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Catheter (N=36) | Standard Catheter (N=36)
Burning in the urethra (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less